CLINICAL TRIAL: NCT00267839
Title: Effects of Exercise on Multiple Risk Factors and Health Costs in Community Living Elderly Women. The Senior Fitness and Prevention Study (SEFIP)
Brief Title: Effect of Exercise on Risk-factors of Elderly Women
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Behinderten- und Versehrten-Sportverband Bayern e.V. (Other); Netzwerk Knochengesundheit e.V. (Unknown); Kassenärztliche Vereinigung Bayern (Unknown); Siemens-Betriebskrankenkasse (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D-ER-OFZ-200501
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Atrophy
Keywords: exercise; intervention; elderly woman; risk factors; health costs; Osteoporosis; cardiovascular diseases; diabetes; Higher Age
MeSH Terms: conditions — Atrophy; Motor Activity; Osteoporosis; Cardiovascular Diseases; Diabetes Mellitus | interventions — Exercise; Health

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Behavioral: physical exercise, wellness

SUMMARY:
The purpose of this study is to determine whether exercise training may impact relevant risk factors and health costs of community living women older 65 years.

DETAILED DESCRIPTION:
The human aging process is associated with a significant increase of risk factors (i.e. osteoporosis, coronary heard disease, diabetes) and a decline in neuromuscular function impacting independence of the subject. Osteoporosis, diabetes type II and arteriosclerosis are diseases known to correlate with age. Participating in regular sport activities elicits numerous favorable effects that contribute to "healthy aging". Unfortunately all existing studies which focus on specific diseases or conditions favour dedicated exercise regimes. However, the complex risk factor scenario of older adults requires multi-purpose exercise programs with impact on all relevant risks. Furthermore so far no exercise study longitudinally determines the effect of an ambulatory exercise program on health cost considering the specific health policy framework of Germany. We hypothesize that regular exercise

1. significantly impact relevant osteoporosis, cardiovascular diseases and diabetes risk factors in elderly subjects
2. significantly reduces health costs in elderly community living women

ELIGIBILITY:
Inclusion Criteria:

* Community living Caucasian woman ≥ 65 years; live expectation > 2 years

Exclusion Criteria:

* secondary osteoporosis
* CVD-events including stroke
* Participation in other studies
* Medication with impact on bone during the last 2 years:

  * bisphosphonates
  * parathormone
  * strontium
  * HRT, anabolic steroids
  * calcitonin
  * natriumflourides
  * active Vit-D-metabolites
  * cortisone > 5 mg/d
* medication with impact on falls
* low physical performance (<50 Watt during ergometry)
* excessive alcohol-intake

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 246 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
health costs after 18 months | baseline 18 month control
falls after 18 months | daily records, analysis after 18 months
Bone parameters after 6, 12 and 18 months | baseline, 6, 12, 18 month-control

SECONDARY OUTCOMES:
Functional status after 6, 12, and 18 months
CHD- and diabetes-risk-factors (bodyfat, blood lipids, glucose, blood pressure) after 6, 12 and 18 months
Quality of live after 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Willi A Kalender, PhD, Study Chair — University of Erlangen-Nürnberg Medical School
Locations (2):
- Germany (2):
  - Institute of Medical Physics University of Erlangen-Nurnberg, Erlangen
  - Institute of Medical Physics, Erlangen

REFERENCES:
- [Background] Kemmler W, von Stengel S, Weineck J, Lauber D, Kalender W, Engelke K. Exercise effects on menopausal risk factors of early postmenopausal women: 3-yr Erlangen fitness osteoporosis prevention study results. Med Sci Sports Exerc. 2005 Feb;37(2):194-203. doi: 10.1249/01.mss.0000152678.20239.76. PMID 15692313
- [Derived] Kemmler W, von Stengel S, Engelke K, Haberle L, Mayhew JL, Kalender WA. Exercise, body composition, and functional ability: a randomized controlled trial. Am J Prev Med. 2010 Mar;38(3):279-87. doi: 10.1016/j.amepre.2009.10.042. PMID 20171529
- [Derived] Kemmler W, von Stengel S, Engelke K, Haberle L, Kalender WA. Exercise effects on bone mineral density, falls, coronary risk factors, and health care costs in older women: the randomized controlled senior fitness and prevention (SEFIP) study. Arch Intern Med. 2010 Jan 25;170(2):179-85. doi: 10.1001/archinternmed.2009.499. PMID 20101013
- See also: Related Info — http://www.imp.uni-erlangen.de